CLINICAL TRIAL: NCT07026071
Title: Effects Of Positional Release Technique Versus Stretching Exercises Combined With Standard Physical Therapy Treatment On Pain, Range Of Motion And Disability In Patients With Chronic Non-Specific Lowback Pain
Brief Title: Positional Release Technique Versus Stretching Exercises In Patients With Chronic Non-Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Burhan- REC/RCR&AHS 24/0140
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Positional Release Technique; Range of Motion; Stretching Exercises
MeSH Terms: conditions — Low Back Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Positional Release Technique
- Group B (Active Comparator)
  Interventions: Other: Stretching Exercises

INTERVENTIONS:
Other: Positional Release Technique — Positional Release Technique will be repeated 3 times in each session for each muscle with an aim to produce a decrease in perceived pain and an increase in pressure tolerance Iliopsoas Quadratus Lumborum Hamstrings
  Arms: Group A
Other: Stretching Exercises — These exercises will be performed with three repetitions per set, three sets per visit and with 30 seconds hold and 30 seconds rest Iliopsoas Quadratus Lumborum Hamstrings
  Arms: Group B

SUMMARY:
This study will be a Randomized Clinical Trial and will be conducted in Physiotherapy Outpatient Department of Allama Iqbal Memorial Teaching Hospital, Sialkot. Non-Probability Convenient Sampling will be used to collect the data. Sample size of subjects with age group between 18-45 years will be taken. Data will be collected from the patients having present complaint of Chronic Non-Specific Low Back Pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Oswestry Disability Index for Disability and Inclinometer for Range of motion. An informed consent will be taken from the participants. Subjects will be selected on the basis of inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive Transcutaneous Electrical Nerve Stimulation, Hot Pack, and Standard Physical Therapy exercises for CNSLBP, while Group A will receive Positional Release Technique for Iliopsoas, Quadratus Lumborum and Hamstring Muscle and Group B will receive Stretching Exercises of Iliopsoas, Quadratus Lumborum and Hamstring Muscle. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

DETAILED DESCRIPTION:
Low back pain (LBP) is considered one of the most prevalent and debilitating musculoskeletal conditions that affects the majority of the general population. It is the most commonly reported complaint area in musculoskeletal conditions, leading to pain and a reduction in overall life quality. Low back pain is pain in the region between the 12th rib and the inferior gluteal fold and is a musculoskeletal system problem that is common in society, mostly caused by nonspecific causes and leads to disability.

Low Back Pain is present in developed countries as well as developing ones, but presents different issues in both: in developed countries, the impact and burden of Non-Specific Low Back Pain is placed on the healthcare and social system first. In contrast, in developing countries, the burden is predominantly placed on the people impacted by low back pain and their support systems.

Nonspecific low back pain is defined as the pain where no specific pathoanatomical cause can be identified and is the most common type of low back pain. A total of 90% of low back pain lacks identifiable pathology and is termed 'non-specific' low back pain (NSLBP). Depending on the duration of the pain, acute low back pain is defined as the pain persisting for less than 06 weeks, Sub-acute Non Specific Low Back Pain refers to pain that lasts between six weeks and three months and chronic non-specific low back pain is the pain when it lasts for more than 12 weeks. Low back pain often becomes chronic, and if non-specific low back pain lasts more than 3 months, it is called chronic non-specific low back pain. Many people with low back pain will experience resolution within 6 weeks of onset. However, two-thirds of people with low back pain report pain at 3 months and 12 months.

Chronic Low Back Pain is a widespread issue that affects many people's daily lives and work abilities. This research compares the Positional Release Technique and Stretching Exercises with standard physical therapy to see which treatment better reduces pain, improves range of motion and decreases disability. The goal of this research is to provide physical therapists with clear evidence on the most effective treatment for CNSLBP, focusing on Iliopsoas, Quadratus Lumborum and Hamstrings Muscle. By identifying the best techniques, this study aims to equip physical therapists with new methods to enhance patient care which, in turn, will aid the healthcare system in providing more effective care.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Gender
* 18 - 45 years of age
* Back Pain with the duration longer than 12 weeks.
* Numeric Rating Scale (NRS) score of 3-7/10
* Oswestry Disability Index score of 20-60
* Minimum 20 degrees of flexion at knee while performing active knee extension test
* Positive Modified Thomas Test
* Participations with Lumbar Pain and Pain in the attachments of Quadratus Lumborum Muscle (iliac crest and lower ribs) or pain localized para spinally or restriction in motion of lumbar due to tightness of Quadratus Lumborum Muscle

Exclusion Criteria:

* Serious spinal disorders, such as fractures
* History of trauma or Previous Spinal Surgery
* Spine osteoarthritis, Spinal Canal Stenosis and Spondylolistheses
* Any neurological symptoms involving Prolapsed Intervertebral Disc, Radiculopathy or presence of root symptoms (e.g. Sciatica and Cauda Equina Syndrome)
* Any systemic disease like Rheumatoid Arthritis, Ankylosing Spondylitis
* Pregnancy, Cancer or Malignancy
* Altered Sensation and Deep Tendon Reflex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
NPRS | Baseline, 4th Week
  PRS stands for Numeric Pain Rating Scale. It's a tool used to measure the intensity of pain, where individuals rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable).
Oswestry Disability Index | Baseline, 4th Week
  The Oswestry Disability Index (ODI) is scored out of 100%, with a lower percentage indicating less disability. The ODI consists of 10 sections, each with 6 statements, scored from 0 to 5, with 0 representing no disability and 5 representing the maximum disability. To calculate the ODI score, sum the scores from all sections, divide by the total possible score (50 if all sections are completed), and multiply by 100.
Lumbar Range of Motion | Baseline, 4th Week
  Lumbar range of motion (ROM) is typically measured in degrees using a goniometer, with normal ranges varying by movement. Flexion is typically around 60-75 degrees, extension 25-35 degrees, and lateral flexion 20-25 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sheeran L, Al-Amri M, Sparkes V, Davies JL. Assessment of Spinal and Pelvic Kinematics Using Inertial Measurement Units in Clinical Subgroups of Persistent Non-Specific Low Back Pain. Sensors (Basel). 2024 Mar 26;24(7):2127. doi: 10.3390/s24072127. PMID 38610338
- [Background] Robinault L, Niazi IK, Kumari N, Amjad I, Menard V, Haavik H. Non-Specific Low Back Pain: An Inductive Exploratory Analysis through Factor Analysis and Deep Learning for Better Clustering. Brain Sci. 2023 Jun 13;13(6):946. doi: 10.3390/brainsci13060946. PMID 37371424
- [Background] Vatovec R, Voglar M. Changes of trunk muscle stiffness in individuals with low back pain: a systematic review with meta-analysis. BMC Musculoskelet Disord. 2024 Feb 19;25(1):155. doi: 10.1186/s12891-024-07241-3. PMID 38373986